CLINICAL TRIAL: NCT00123240
Title: High Carbohydrate vs. High Fat Diets in the Treatment of Obesity (JBR 0512)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBR-0512
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Obesity
Keywords: overweight; obese; diet
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Fat/Protein Diet (Active Comparator)
  Interventions: Behavioral: Low calorie high fat/protein diet
- High Carbohydrate Diet (Active Comparator)
  Interventions: Behavioral: Low calorie high carbohydrate diet

INTERVENTIONS:
Behavioral: Low calorie high carbohydrate diet — 65% carbohydrate, 15% protein, 20% fat (7% SFA, 8% MFA, 4% PUFA), P/S 0.63, 152 mg cholesterol/1500 kcal
  Arms: High Carbohydrate Diet
Behavioral: Low calorie high fat/protein diet — High Fat/Protein Diet: 10% carbohydrate, 25% protein, 65% fat (26% SFA, 25% MFA, 9% PUFA), P/S 0.33, 458 mg cholesterol/1500 kcal
  Arms: High Fat/Protein Diet

SUMMARY:
The purpose of this study is to compare the ability of low calorie high carbohydrate and low calorie high fat/protein diets to decrease abdominal fat in overweight and obese subjects. The investigators will also test the effects of these diets on secondary outcomes including body composition, fluid and electrolyte balance, lipids and lipoproteins, blood pressure, arterial compliance, glucose and insulin metabolism, bone turnover, and measures of satiety.

DETAILED DESCRIPTION:
Participation in this study requires 2 screening visits to the outpatient clinic, and if participants qualify, 10 inpatient study weeks.

Subjects will be admitted to the Rockefeller University Hospital for the 10 week in-patient phase of the study. The first 2 weeks consist of a weight stabilization period, during which subjects will be required to consume an average American diet. This is followed by the 6 week weight loss period where subjects will be randomized to either a low calorie high carbohydrate or a low calorie high fat/protein diet. On both diets there will be a 50% calorie deficit compared to the weight stabilization period. This will be followed by a 2 week weight maintenance period during which calories will be added to the diet to maintain the new weight. Appropriate adjustments will be made to keep the subject's weight stable.

During the entire inpatient study, subjects will consume one multivitamin per day (Centrum, always complete, from A to Zinc) and one iron supplement per day. In addition, unlimited access to zero calorie liquids (water/diet soda) will be available and will be encouraged to maintain one's usual activity level.

Females of reproductive age, need to make sure that they do not become pregnant during the inpatient study. Urine will be tested for pregnancy once during the stabilization and weight maintenance phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Man or a woman with a body mass index (BMI) of 30 to 34.9
* Man with a BMI of 25 to 29.9 with a waist circumference > 102cm (40in)
* Woman with a BMI of 25 to 29.9 with a waist circumference > 88cm (35in)

Exclusion Criteria:

* High Blood Pressure
* High Cholesterol
* Diabetes
* HIV positive
* Syphilis
* Hepatitis B/C positive

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Visceral adipose tissue | days 12, 68

SECONDARY OUTCOMES:
Body composition | days 12, 68
Blood pressure | days 11 and 67
Insulin glucose metabolism | days 13, 15 69, 71
Bone turnover | days 14, 70
Measures of satiety | once a week

CONTACTS AND LOCATIONS:
Overall Officials: Jan L. Breslow, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.rucares.org